CLINICAL TRIAL: NCT07246954
Title: A Chaplain-clinician Led Spiritual Care (PEACE) Intervention on Spiritual/Religious Beliefs Related to Medical Care in Patients With Advanced Cancer: a Pilot Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-1052; NCI-2025-08254 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-11-04; First posted 2025-11-24 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Spiritual Care; Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): Patients will participate in two PEACE intervention sessions, which will last 30-60 minutes each.
  Interventions: Other: Peace Intervention
- Phase 2 (Experimental): Usual care is a comprehensive evaluation of the physical, emotional, and spiritual needs of the patient by the Supportive/Palliative Care medical team
  Interventions: Other: Peace Intervention; Other: Usual Care

INTERVENTIONS:
Other: Peace Intervention — Patients will participate in two PEACE intervention sessions, which will last 30-60 minutes each.
Other: Usual Care — Usual care is a comprehensive evaluation of the physical, emotional, and spiritual needs of the patient by the Supportive/Palliative Care medical team.
  Arms: Phase 2

SUMMARY:
To examine the feasibility and acceptability of chaplain-clinician led spiritual care (PEACE: Perception, Exploring, Addressing, Compassionate Connection, Embracing) intervention in patients with advanced cancer.

DETAILED DESCRIPTION:
Primary Objectives

(Phase 1): To examine the feasibility and acceptability of a Chaplain-Clinician led spiritual care (PEACE: Perception, Exploring, Addressing, Compassionate Connection, Embracing) intervention in patients with advanced cancer admitted to a comprehensive cancer center in a single-arm pilot trial. Evaluation of feasibility will be per ≥70% participation in all sessions.

Acceptability will be assessed as ≥70% reporting satisfaction and ≥70% recommending PEACE intervention to others at the post-treatment assessment.

(Phase 2): To examine the within-group change in the influence of spiritual/religious beliefs on medical care (Question 2 in the Religious Beliefs in End-of-Life Medical Care [RBEC] tool: I will accept every possible medical treatment because my faith tells me to do everything I can to stay alive longer) from baseline to post-intervention assessments at 2 + 1 days in participants who participate in the PEACE intervention group and the usual care group.

ELIGIBILITY:
Eligibility Criteria

1. Participants with advanced cancer (locally advanced, metastatic, recurrent, or incurable) seen by the participant supportive/palliative care mobile team at MD Anderson Cancer Center.
2. Respond "somewhat to A great deal" to the question in the RBEC questionnaire "I will accept every possible medical treatment because my faith tells me to do everything I can to stay alive longer".
3. Participant s aged 18 years or over.
4. Karnofsky performance status ≥30% at time of inclusion into study.
5. Normal cognitive status as determined by the supportive care clinicians based on the ability to understand the nature of the study and consent process.
6. Only English-speaking, as determined by their ability to understand the informed consent, the intervention, and the assessment tools.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
RBEC Questionnaire | Through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Delgado Guay, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org